CLINICAL TRIAL: NCT02422134
Title: Novel Approach for Embryo Transfer Medium by Adding Cytokine to Hyaluronan Enriched Embryo Transfer Medium (Embryo Glue)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banon IVF Center Assiut, Egypt (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Ibnsina IVF Sohag
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Infertility
Keywords: Pregnancy; implantation; Cytokine
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cytokine plus Hyalurinan embryo transfer arm (Active Comparator): To monitor the pregnancy and implantation of the patients in this arm after adding Cytokine to the embryo transfer medium.
  Interventions: Other: Cytokine group
- Hyalurinan embryo transfer group (No Intervention): To transfer the embryos using a Hyaluronan enriched medium only

INTERVENTIONS:
Other: Cytokine group — Testing the efficacy of adding Cytokine to embryo transfer medium
  Arms: Cytokine plus Hyalurinan embryo transfer arm

SUMMARY:
It was proven that the Cytokine granulocyte-Macrophage clony stimulating factor had been found naturally in reproductive tract so our target is to test its effect if added to embryo transfer medium.

DETAILED DESCRIPTION:
The IVF embryo transfer media design and upgrade underwent many ideas during the last 3 decades, we suppose that adding Cytokine GM-CSF as an endometrial modifier to already proven successful medium hyaluronan enriched medium to test the efficacy ipon pregnancy and implantation rate in vitro so we decide to design a trial to compare the clinical outcome by sibling embryo to be transferred into 2 groups and the same culture condition but with one arm with Cytokine and the other is traditional one and closely monitor the outcome within the 2 arms and record the results.

ELIGIBILITY:
Inclusion Criteria:

* all patients

Exclusion Criteria:

* above 40 years old

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate ( % ) | 9 months

SECONDARY OUTCOMES:
Implantation rate ( % ) | 9 months

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Banon IVF center, Asyut
  - Ibnsina IVF center, Sohag